CLINICAL TRIAL: NCT04426994
Title: Hypomagnesemia Associated With Proton-Pump Inhibitor Use
Acronym: PPI_HypoMg
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PPI HypoMg
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Proton Pump Inhibitor Adverse Reaction; Hypomagnesemia; Arrhythmias, Cardiac; Seizures; Hypocalcemia; Hypokalemia
MeSH Terms: conditions — Arrhythmias, Cardiac; Seizures; Hypocalcemia; Hypokalemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: Patients admitted with hypomagnesemia are evaluated for proton pump inhibitor use and likelihood of hypomagnesemia due to proton pump inhibitor use
  Interventions: Drug: proton pump inhibitor use
- Control: Patients on long-term proton pump inhibitor without documented hypomagnesemia
  Interventions: Drug: proton pump inhibitor use

INTERVENTIONS:
Drug: proton pump inhibitor use — Patients using long term proton pump inhibitor

SUMMARY:
Use of proton pump inhibitors has been associated with hypomagnesemia. However, various case-control or prospective studies have found conflicting results with regards to proton pump inhibitors use and development of hypomagnesemia. Our aim was to evaluate the likelihood that proton pump inhibitors contributed to severe hypomagnesemia in a retrospective cohort of patients admitted with severe hypomagenesemia. We also aimed to look for risk factors leading to development of hypomagnesemia amongst users of proton pump inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with hypomagnesemia (cases)
* Patients prescribed with proton pump inhibitors (controls)

Exclusion Criteria:

* Patients prescribed with less than three months duration of proton pump inhibitors (controls)

Ages: 14 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients managed at a referral centre from 2013 - 2016. Cases were admitted to the referral centre and had documentation hypomagnesemia. Controls were prescribed a course of proton pump inhibitor during the same period
Sampling Method: Probability Sample
Enrollment: 211672 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Hypomagnesemia due to use with proton pump inhibitor | 2013 to 2016
  Number of patients with Hypomagnesemia related to use of proton pump inhibitor using Naranjo score

SECONDARY OUTCOMES:
Risk factors for Hypomagnesemia | 2013 to 2016
  Odds ratio of developing Hypomagnesemia with risk factors of age, gender, type of drug, dose of drug, chronic renal failure, use of diuretics
Hypocalcaemia | 2013 to 2016
  Number of patients developing hypocalcemia
Hypokalemia | 2013 to 2016
  Number of patients developing Hypokalemia

CONTACTS AND LOCATIONS:
Overall Officials: Troy H Puar, MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised pooled data